CLINICAL TRIAL: NCT04353349
Title: Impact of Minimally Invasive Robotic Approach Compared to VATS and Open Approach on Quality of Life and Immune Response in Patients Candidated to Lobectomy or Anatomical Segmentectomy
Brief Title: Impact of Robotic Approach Compared to VATS and Open Approach on Quality of Life in Patients With Lung Cancer
Acronym: QoL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1524
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Robotic Thoracic Surgery; Video-assisted Thoracis Surgery (VATS); Open Thoracotomy Surgery
Keywords: Robotic surgery; Lung cancer; Early stage; Quality of life; Post-operative pain
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients operated with an open approach
- Patients operated with minimally invasive robotic approach
- Patients operated with VATS approach

SUMMARY:
The aim of the study is to compare quality of life and early and late post-operative pain after anatomical lung resection (lobectomy or segmentectomy) performed by a robotic approach compared to the videothoracoscopic approach (VATS) and the thoracotomic approach antero-lateral in patients with early stage lung cancer.

ELIGIBILITY:
Inclusion Criteria :

* known or suspected lung cancer clinical stage T1-T2;
* N0-N1 candidates for surgery lobectomy or anatomical segmentectomy;
* ASA-1-2-3;
* not severe heart disease;
* no alcohol;
* no renal impairment (creatinine <2);
* not obese (BMI <30);
* no evidence of other serious comorbidities in the opinion of the investigator.

Exclusion Criteria:

* severe heart disease;
* renal impairment (creatinine >2.5);
* evidence of any serious comorbidities according to the investigator;
* malignant tumor in the previous 2 years;
* previous chest surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population should have the following Inclusion criteria: - known or suspected lung cancer clinical stage T1-T2, N0-N1 candidates for surgery lobectomy or anatomical segmentectomy; - ASA-1-2-3; - not severe heart disease; -no alcohol; -no renal impairment (creatinine <2); -not obese (BMI <30); no evidence of other serious comorbidities in the opinion of the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life by EORTC QOL-CC30. | 01/04/2016 - 01/12/2020
  The sample size is calculated on the primary end point which is the prospective evaluation of quality of life (QoL) evolution after robotic-assisted thoracoscopic resection versus videothoracoscopic resection versus
  open thoracotomy, with the European Organisation for Research and Treatment of Cancer (EORTC) QoL Questionnaire-C30 and the lung cancer-specific module, LC-13.
  51 patients operated in each group will provide 80% power to detect a 8-point difference in mean QLQ-C30 "Pain score" between any two study groups, at the 5% level of significance assuming a coefficient of variability of 0.5 and using a two-sided two-sample t-test. The scale parameters range are included from 1 (not at all) to 4 (very much).

SECONDARY OUTCOMES:
Evaluation of postoperative pain by daily evaluation with visual numeric scale before and after surgery until discharge and at 1, 6 and 12 months | 01/04/2016 - 01/12/2020
  Pain assessment will be recorded daily starting from the pre-operative day and post-operatively until discharge and subsequently at 2 weeks, 6 months and 12 months after surgery with numerical scale from 0 to 10 (ENV pain score); via questionnaire "Brief Pain Inventory".
  A value of ENV ≤3 will be attributed to adequate analgesia; ENV a score of 4 to 6 will be considered inadequate analgesia with administration of analgesia as needed; ENV score ≥7 will be considered poor analgesia.
Intraoperative complications | 01/04/2016 - 01/12/2020
  Conversion rate, defined as procedures that start with minimally invasive access and are converted to open surgery due to different reasons (bleeding, anatomical reasons, oncological reasons, technical reasons, other).
Postoperative complications | 01/04/2016 - 01/12/2020
  Surgical complications, higher or equal grade II assessed by Clavien-Dindo scale, within 90 days.
Disease free survival at 24 months | 01/04/2016 - 01/12/2020
  Disease free survival will be explored with survival analysis. The time will be calculated from the surgery data to the first recurrence date or to last contact date for all the patients free of disease at the end of surgery. Difference between groups will be explored with log-rank test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy